CLINICAL TRIAL: NCT01008293
Title: Health Related Quality of Life in Patient With Chronic Liver Disease and Effect of Probiotics in the Treatment of MHE and Health Related Quality of Life
Brief Title: Effect of Probiotics in Treatment of Minimal Hepatic Encephalopathy (MHE) and Health Related Quality of Life
Acronym: MHE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: CD Pharma India Pvt. Ltd. (Industry)
Collaborators: Indian Council of Medical Research (Other Government); All India Institute of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MHE-VSL3-YKJ_AIIMS_ver1
Record Dates: First submitted 2009-11-04; First posted 2009-11-05 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Chronic Liver Disease; Hepatic Encephalopathy
MeSH Terms: conditions — Hepatic Encephalopathy | interventions — Lactulose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- VSL#3 (Experimental)
  Interventions: Drug: VSL#3
- Lactulose (Active Comparator): 30-60 ml of lactulose per day (2 months) to ensure 2-3 soft stools
  Interventions: Drug: Lactulose

INTERVENTIONS:
Drug: VSL#3 — VSL#3 (2 capsules bid.for 2 months, Each containing 112.5 billion viable lyophilized bacteria). Each capsule contains 4 strains of Lactobacillus (L. casei, L. plantarum, L. acidophilus, and L. delbrueckii subsp. bulgaricus), 3 strains of Bifidobacterium (B. longum, L. breve, and B. infantis), and 1 strain of Streptococcus salivarius subsp. thermophilus (designated hereafter as S. thermophilus)
  Arms: VSL#3
Drug: Lactulose — 30-60 ml of lactulose per day for 2 months to ensure 2-3 soft stools.
  Other Names: Duphalac
  Arms: Lactulose

SUMMARY:
This study is a randomized, open, parallel group, active comparator, single center trial. Objectives of the study are hereby given below:

* To study the health related quality of life (HRQOL) in patients with chronic liver disease.
* To assess the prevalence of minimal hepatic encephalopathy (MHE) in patients with chronic liver disease and assessment of HRQOL in patients with MHE.
* To compare the effect of probiotics and lactulose in the treatment of MHE
* To assess the effect of probiotics and lactulose on the HRQOL in patients with MHE.

DETAILED DESCRIPTION:
The study design would comprise of two parts

1. Part I: Cross sectional study: This part would comprise of the assessment of HRQOL in patients with CLD

   1. All the consecutive patients diagnosed as CLD would be enrolled in the study. All these patients would be enrolled from the liver clinics of the department of gastroenterology and those admitted in the gastroenterology ward at AIIMS.
   2. Alcohol would be considered to be the cause of CLD, if the patient regularly consumed ≥80g/d of alcohol for five years
   3. The staging of cirrhosis would be done according to the Child Pugh classification: A, B and C
   4. The causes of CLD would be divided into:- viral hepatitis, alcohol, viral hepatitis combining with alcohol and miscellaneous causes
2. Part II: Prospective randomized controlled trial: In this part the outcome of lactulose and probiotic therapy in the treatment of MHE and its effect on the HRQOL will be compared.

   1. All the consecutive patients with CLD without overt encephalopathy would be screened for MHE.
   2. All these patients would be enrolled from the liver clinics and the gastroenterology ward, AIIMS.
   3. The diagnosis of MHE would be based on abnormal psychometric tests (NCT-A and NCT-B or FCT-A and FCT-B) and /or abnormal P300 auditory event related potentials.

ELIGIBILITY:
Inclusion Criteria:

* All the patients with Chronic Liver Disease or Minimal Hepatic Encephalopathy (without overt hepatic encephalopathy) aged between 15 to 80 years of both the genders would be enrolled consecutively.

Exclusion Criteria:

* Patients with overt hepatic encephalopathy
* Active medical co-morbidities like CHD, chronic respiratory disease, chronic renal disease, malignancies, diabetes etc
* Malignancy
* History of taking lactulose or probiotics or antibiotics, in the past 6 weeks
* Presence of other neurological or psychiatric disorder
* Patients who underwent shunt surgery for portal hypertension
* History of taking medicines likely to interfere with psychometric performance
* History of GI hemorrhage or spontaneous bacterial peritonitis during the past 6 weeks
* Presence of mature cataracts and diabetic retinopathy
* Refused to participate in the study

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-10; Primary Completion 2012-06 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
To compare the effect of probiotics and lactulose based on normalization of the abnormal test parameters, Neuropsychometric tests, P3ERP, EEG, venous ammonia levels, Development of overt encephalopathy and other complications and HRQOL | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Y K Joshi, Prof., Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- Dept. of Gastroenterology and H.N.U., All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India